CLINICAL TRIAL: NCT01511445
Title: Interbody Fusion Devices in the Treatment of Cervicobrachial Syndrome; a Blinded Randomised Trial of Cancellous Structured Ceramic (CSC) Versus PEEK Cages.
Brief Title: Interbody Fusion Devices in the Treatment of Cervicobrachial Syndrome
Acronym: CASCADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amedica Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Amedica 2010-1; NL36103.098.11 (Registry Identifier: Netherlands Trial Registry)
Record Dates: First submitted 2012-01-13; First posted 2012-01-18 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Radiating Pain; Myelopathy; Cervicobrachial Syndrome
Keywords: Cervicobrachial pain; radicular pain; arm pain; myelopathy; radiculitis; Radiating pain with or without signs of myelopathy.
MeSH Terms: conditions — Pain; Spinal Cord Diseases; Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACDF with PEEK interbody cage (Active Comparator): Anterior cervical discectomy and fusion (ACDF) with an interbody spacer made from polyetheretherketone (PEEK) plastic. The open space in the center of the cage is to be filled with local autologous bone harvested during the decompression phase of the procedure.
  Interventions: Device: Anterior cervical discectomy and fusion (ACDF) with PEEK Cage
- ACDF with Valeo CSC Ceramic Cage (Experimental): ACDF with the Valeo CSC cage, a silicon nitride ceramic interbody cage. The center area of the cage is filled with porous silicon nitride. No autologous bone is used; the cage is soaked in patient blood.
  Interventions: Device: Anterior cervical discectomy and fusion (ACDF) with a Valeo CSC Cage

INTERVENTIONS:
Device: Anterior cervical discectomy and fusion (ACDF) with PEEK Cage — Anterior cervical discectomy and fusion with the use of a PEEK plastic interbody spacer
  Other Names: Medicrea Manta or similar PEEK cage
  Arms: ACDF with PEEK interbody cage
Device: Anterior cervical discectomy and fusion (ACDF) with a Valeo CSC Cage — Anterior cervical discectomy and fusion with a Valeo ceramic cage interbody spacer.
  Other Names: Valeo CSC (Cancellous Structured Ceramic); Silicon Nitride ceramic
  Arms: ACDF with Valeo CSC Ceramic Cage

SUMMARY:
This study randomizes neck and arm pain patients being treated with discectomy and anterior interbody fusion into two groups: one to receive a new ceramic implant and a control group with a more traditional plastic implant. The study will measure and compare pain and disability improvement with the two products over a period of two years. The fusion status will also be judged with plane x-rays and one CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 75 years
* Radicular signs and symptoms in one or both arms (i.e., pain, paraesthesiae or paresis in a specific nerve root distribution) or symptoms and signs of acute or chronic myelopathy.
* At least 8 weeks prior conservative treatment (i.e., physical therapy, pain medication)
* Radiographic diagnosis of cervical disc herniation and/or osteophyte at 1 level (C3-C4 to C7-T1) in accordance with clinical signs and symptoms
* Ability and willingness to comply with project requirements
* Written informed consent given by the subject or the subject's legally authorised representative

Exclusion Criteria:

* Previous cervical surgery (either anterior or posterior)
* Increased motion on dynamic studies (> 3 mm)
* Severe segmental kyphosis of the involved disc level (> 7 degrees)
* Patient cannot be imaged with MRI
* Neck pain only (without radicular or medullary symptoms)
* Infection
* Metabolic and bone diseases (osteoporosis, severe osteopenia)
* Neoplasma or trauma of the cervical spine
* Spinal anomaly (Klippel Feil, Bechterew, OPLL)
* Severe mental or psychiatric disorder
* Inadequate Dutch language
* Planned (e)migration abroad in the year after inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Arts, MD, PhD, Principal Investigator — Medical Center Haaglanden
Locations (1):
- Medical Center Haaglanden, The Hague, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed as double-blind randomized trial. The design called for randomizing 100 patients.
Pre-assignment Details: Four additional patients were randomized when four patients were excluded for protocol violations prior to the primary endpoint. A surgeon who had not been trained as an investigator operated on these four patients, making numerous protocol violations in implant technique. These patients were randomized and had pre-op data in the study.
Period: Overall Study
Arm/Group | ACDF With Valeo CSC Ceramic Cage | ACDF With PEEK Interbody Cage
Started (Enrollment) | 53 (Patient enrollment started in December, 2011.) | 51 (Patient enrollment started in December, 2011.)
Surgeries Completed | 53 (All surgeries were completed by October, 2013.) | 51 (All surgeries were completed by October, 2013.)
Primary Completion October, 2014 | 48 (1 was excluded Bechterew's disease. 1 protocol violation. 3 were lost to follow-up.) | 47 (3 protocol violations. 1 lost to follow-up.)
Follow-up Completion | 48 (Two year follow-up was completed in November, 2015) | 47 (Two year follow-up was completed in November, 2015)
Completed | 48 (Data analysis was completed in February, 2016) | 47 (Data analysis was completed in February, 2016)
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ACDF With Valeo CSC Ceramic Cage: ACDF with the Valeo CSC cage, a silicon nitride ceramic interbody cage.
- ACDF With PEEK Interbody Cage: Anterior cervical discectomy and fusion (ACDF) with an interbody spacer made from polyetheretherketone (PEEK) plastic.
- Total: Total of all reporting groups
Arm/Group | ACDF With Valeo CSC Ceramic Cage | ACDF With PEEK Interbody Cage | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at date of surgery
  years | 53.3 (9.3) | 49.6 (9.5) | 51.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 26 | 26 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 53 | 51 | 104
Use of nicotine products [Count of Participants; unit: Participants] | 23 | 20 | 43
Symptomatic (operated) spinal level [Count of Participants; unit: Participants] — Patients were operated at a single cervical spinal level from C3-C4 to C7-T1
  Participants
    C3-C4 | 1 | 1 | 2
    C4-C5 | 0 | 6 | 6
    C5-C6 | 30 | 30 | 60
    C6-C7 | 20 | 12 | 32
    C7-T1 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Neck Disability Index
Description: The change in the Neck Disability Index compared to the pre-op value for each group will be compared. Neck disability index is a unitless measure from zero (no disability) to 100 (absolute disability). Change is calculated as the pre-op value minus the 24 month value. A negative difference indicates that the patient is more disabled at 24 months.
Time Frame: 24 months post-op
Population: Patients who had data from 24 month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 100
Arm/Group | ACDF With Valeo CSC Ceramic Cage | ACDF With PEEK Interbody Cage
Number analyzed (Participants) | 47 | 44
units on a scale from 0 to 100 | 17.9 (14.9) | 16.7 (16.1)
Statistical Analysis 1: Comparison: ACDF With Valeo CSC Ceramic Cage vs ACDF With PEEK Interbody Cage; The null hypothesis was that the mean change in NDI scores from pre-op to 24 months was equal in the two study arms; Test type: Non-Inferiority — The noninferiority margin was specified as 15 NDI points (0-100 scale); p = 0.641, Fisher Exact; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-7.3 to 4.5], Standard Error of Mean 2.96 — A negative value means that the PEEK change was slightly larger than the silicon nitride study arm

2. Secondary Outcome: Fusion Status
Description: Dynamic flexion-extension plane film x-rays will be used to assess fusion at all four follow-up periods. The criteria for fusion are rotation motion less than or equal to four degrees and translation less than 1.25 mm. The final fusion judgement will be fusion status at 24 months or the last time point with flexion-extension data available.
Time Frame: 3 mo., 6mo., 12 mo., 24 months
Population: Patients with 24 month films
Measure: Count of Participants; unit: Participants
Arm/Group | ACDF With Valeo CSC Ceramic Cage | ACDF With PEEK Interbody Cage
Number analyzed (Participants) | 43 | 41
Participants | 40 | 37
Statistical Analysis 1: Comparison: ACDF With Valeo CSC Ceramic Cage vs ACDF With PEEK Interbody Cage; The null hypothesis was that the fusion rates would be equal in the two study arms. The comparison includes patients with flexion-extension films at 24 months (as-treated population); Test type: Non-Inferiority — The definition of fusion is rotation on flexion-extension films of less than or equal to four degrees and translation less than 1.25 mm; p = 0.710, Fisher Exact

ADVERSE EVENTS:
Description: Investigators completed adverse event questionnaires and patients were surveyed for adverse events at each interaction with the investigational team
Arm/Group | ACDF With Valeo CSC Ceramic Cage | ACDF With PEEK Interbody Cage
Serious Adverse Events (participants affected / at risk) | 2/53 | 1/51
Other Adverse Events (participants affected / at risk) | 16/53 | 11/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACDF With Valeo CSC Ceramic Cage (N=53) | ACDF With PEEK Interbody Cage (N=51)
Replacement of implant due to subsidence (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Cage subsidence led to symptoms; revised by removing cage and replacing with bone graft and a cervical plate
Debridement of abscess (Infections and infestations) | 1 (1) | 0 (0) — The abscess was cleaned in a second surgery without cage removal
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACDF With Valeo CSC Ceramic Cage (N=53) | ACDF With PEEK Interbody Cage (N=51)
Dysphasia (Injury, poisoning and procedural complications) | 9 (9) | 8 (8) — Difficulty swallowing in the immediate post-op period. All cases resolved completely as post-op swelling subsided.
Surgery at additional spinal level (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) — Surgery for development of new or persistent symptoms. More common at lower cervical spine levels.
Removal for restenosis (Immune system disorders) | 1 (1) | 0 (0) — Patient had undiagnosed Becherew's disease (ankylosing spondylitis), an exclusion criterion for the study. A bone spur regrew underneath the cage. The patient had a revision with bone graft and a cervical plate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No